CLINICAL TRIAL: NCT05518929
Title: The Incidences Of Hypoxia And Severe Hypoxia During Gastroenterological Endoscope Procedures Sedated With Ciprofol Compared With Propofol In Overweight Or Obesity Adults Patients, A Multicenter, Randomized, Controlled Trial
Brief Title: Hypoxia During Gastroenterological Endoscope Procedures Sedated With Ciprofol In Overweight Or Obesity Patients
Acronym: SpO2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Zhejiang Tumor Hospital (Other); Beijing Hospital (Other Government); Second Hospital of Shanxi Medical University (Other); Dalian Municipal Friendship Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2022-155-B
Record Dates: First submitted 2022-08-24; First posted 2022-08-29 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Gastric Ulcer; Gastric Cancer; Gastrointestinal Polyp
Keywords: Ciprofol; Gastroenterological Endoscope; Overweight; Obesity
MeSH Terms: conditions — Stomach Ulcer; Stomach Neoplasms; Overweight; Obesity | interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; Propofol

STUDY DESIGN:
Intervention Model Description: Multicenter, Randomized, Open-label, Propofol-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group(Propofol group) (Active Comparator): Anesthesia induction:Propofol 1.5mg/kg Anesthesia maintenance: Propofol 0.75mg/kg
  Interventions: Drug: Propofol
- Experimental group(ciprofol group) (Experimental): Anesthesia induction:ciprofol 0.4mg/kg Anesthesia maintenance: ciprofol 0.2mg/kg
  Interventions: Drug: Ciprofol

INTERVENTIONS:
Drug: Ciprofol — The sedation of gastrointestinal endoscopy with Ciprofol
  Arms: Experimental group(ciprofol group)
Drug: Propofol — The sedation of gastrointestinal endoscopy with Propofol
  Arms: Control group(Propofol group)

SUMMARY:
Ciprofol is a new general anesthetic, which combine with γ- Aminobutyric acid-a (GABAA) receptor. Ciprofol has shown equivalent anesthetic efficacy of propofol at 1/4 to 1/5 of the dosage. Ciprofol has the pharmacodynamic characteristics of rapid onset, stable and rapid recovery. Phase III clinical results showed that the incidence of injection pain and respiratory and circulatory depression of ciprofol was lower than that of propofol. Therefore, ciprofol has a good application prospect in the sedation for gastrointestinal endoscopy, especially for overweight and obese patients. We conduct a Multicenter, Randomized, Open-label, Propofol-controlled Study to Evaluate the incidence of hypoxia and severe hypoxia during Gastroenterological Endoscope sedated with CiProfol in Overweight or Obesity patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age, ≤18 and ≤80 years, no gender limit
2. Undergoing routine gastrointestinal endoscopic diagnosis and treatment
3. American Society of Aneshesiologists (ASA) classification I-II
4. Body mass index (BMI) ≥ 23kg/m2
5. Estimated procedure duration less than 30 min
6. Clearly understand and voluntarily participate in the study; provide signed informed consent

Exclusion Criteria:

1. Need to perform complicated endoscopic techniques for diagnosis and treatment, such as cholangiopancreatography surgery, endoscopic ultrasonography, endoscopic mucosal resection, endoscopic submucosa stripping, and oral endoscopic muscle dissection
2. Intend to undergo tracheal intubation or laryngeal mask
3. Patients' SpO2 ≤ 95% after entering the endoscope room;
4. Be definitely diagnosed as obstructive sleep apnea hypopnea syndrome;
5. Body weight < 40kg
6. Have serious heart diseases such as severe arrhythmia, heart failure, Adams-Stokes Disease, unstable angina pectoris, myocardial infarction in the last 6 months, history of tachycardia / bradycardia requiring medical treatment, third degree atrioventricular block or QTC interval ≥ 450ms (corrected according to fridericia's formula), or exercise tolerance < 4mets
7. Systolic blood pressure ≥ 180mmhg or / and diastolic blood pressure ≥ 110mmhg measured in the endoscope room
8. Respiratory insufficiency, history of obstructive pulmonary disease, history of bronchospasm requiring treatment within 3 months, acute respiratory tract infection within 1 week, and obvious symptoms such as fever, wheezing, nasal congestion and cough
9. There is an uncontrolled disease history with significant clinical significance, such as liver, kidney, blood system, nervous system or metabolic system, which may not be suitable for participating in the study
10. Pregnant or breast-feeding women
11. Allergy to eggs, soy products, opioids and other drugs, propofol, etc.
12. Participated in other clinical trials as a subject within 3 months
13. Unhealthy alcohol drinking, defined by more than three standard drinks per day (≈10 g alcohol , equivalent to 50 g of strong Chinese spirits)
14. Patients with brain injury, possible convulsion, myoclonus, intracranial hypertension, cerebral aneurysm, cerebrovascular accident history, schizophrenia, intellectual disability, mania, psychosis, long-term use of psychotropic drugs, drug addiction, cognitive dysfunction history, etc.
15. Patients who the investigator considers inappropriate to participate in this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1090 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of hypoxia and severe hypoxia | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  hypoxia( 75%≤SpO2≤89% for<60s);severe hypoxia(SpO2<75%，or SpO2<90% for >60s)

SECONDARY OUTCOMES:
Incidence of hypoxia | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  hypoxia( 75%≤SpO2≤89% for<60s)
Incidence of severe hypoxia | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  severe hypoxemia(SpO2<75%，or SpO2<90% for >60s)
Incidence of subclinical respiratory depression | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  subclinical respiratory depression（90% ≤SpO2 ≤95% ）
Success rate of gastroenteroscopy endoscope | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
Incidence of injection pain when the intravenous administration of Ciprofol or propofol for sedation assessed by questionnaire. | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  Patients complain pain at the site of injection or tell investigators feeling pain when they were asked before they lose consciousness.
Proportion of corrective hypoxic measures | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  Treatment of patients with hypoxia

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, Study Director — Department of Anesthesiology Renji Hospital
Locations (5):
- China (5):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Zhejiang Tumor Hospital, Zhejiang, Hangzhou
  - Dalian Municipal Friendship Hospital, Dalian, Liaoning
  - Renji Hospital, Shanghai, Shanghai Municipality
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou R, Dai W, Su Z, Lian Y, Wen P, Zhang L, Kong L, Hua Z, Sun Y, Zhao H, Wang Q, Yu W, Su D. Ciprofol Versus Propofol for the Prevention of Hypoxia During Gastrointestinal Endoscopy Procedures in Overweight Patients: A Multicenter, Randomized, Controlled Trial. Dig Endosc. 2026 Feb;38(2):e70102. doi: 10.1111/den.70102. PMID 41626789